CLINICAL TRIAL: NCT01380600
Title: A Phase 1b Dose Escalation Study of JX-594 (Thymidine Kinase-Inactivated Vaccinia Virus Plus GM-CSF) Administered by Biweekly (Every Two Weeks) Intravenous Infusion in Patients With Metastatic, Refractory Colorectal Carcinoma
Brief Title: Safety Study of Recombinant Vaccinia Virus Administered Intravenously in Patients With Metastatic, Refractory Colorectal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Sponsor
Organization: SillaJen, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX594-IV-CRC014
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2012-03

CONDITIONS: Carcinoma, Colorectal
Keywords: Vaccinia; Vaccinia Virus; JX-594; Jennerex; Colorectal Carcinoma; Colorectal cancer; Colon Cancer; Rectal Cancer; Pexa-Vec
MeSH Terms: conditions — Colorectal Neoplasms; Vaccinia; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm; Dose escalation (Other): Dose escalation 1e6 pfu/kg bw, 1e7 pfu/kg bw, 3e7 pfu/kg bw of Recombinant Vaccinia GM-CSF JX-594
  Interventions: Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)

INTERVENTIONS:
Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594) — Intravenous Dose Range: 1x10^6 pfu/kg, 1x10^7 pfu/kg, 3x10^7 pfu/kg Up to 4 intravenous infusions administered over 60 minutes every 2 weeks.
  Other Names: JX-594

SUMMARY:
The purpose of this pilot safety study is to evaluate the safety and tolerability of JX-594 (Pexa-Vec) administered intravenously every 2 weeks in colorectal carcinoma patients who are refractory to or intolerant of oxaliplatin, irinotecan, and Erbitux treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, advanced/metastatic colorectal carcinoma
* Failed both oxaliplatin and irinotecan based regimens for advanced/metastatic disease (if tumor advanced either immediately or within 3 months of the end of treatment)
* Resistance to Erbitux: patients with Ras mutations, or for whom Erbitux has failed (if tumor advanced either immediately or within 3 months of the end of treatment, or there is no response to Erbitux therapy due to a lack of expression of EGFR (epidermal growth factor))
* Karnofsky Performance Score (KPS) ≥ 70
* Age ≥18 years
* Laboratory Safety: WBC ≥ 3,500 cells/mm3 and ≤ 50,000 cells/mm3, ANC ≥ 1,500 cells/mm3, Hemoglobin ≥ 10 g/dL (transfusion allowed), Platelet count ≥ 100,000 plts/mm3,Total bilirubin ≤ 1.5 X ULN, INR ≤ 1.5, AST, ALT ≤ 2.5x ULN (in case of liver metastasis: AST,ALT ≤5.0 x ULN)
* Serum chemistries within normal limits (WNL) or Grade 1 (excluding alkaline phosphatase) - If patients are diabetic, a fasting glucose must be done and patients must be > 160 mg/dL.
* Patients who, if they are sexually active, are willing and able to refrain from sexual activity for 3 weeks following JX-594 administration. Patients who are willing and able to use a permitted contraceptive for 3 months after the final administration of JX-594.

Exclusion Criteria:

* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids)
* Known myeloproliferative disorders requiring systemic therapy
* History of exfoliative skin condition (e.g. eczema or ectopic dermatitis) requiring systemic therapy
* History of acquiring opportunistic infections.
* Tumor(s) invading a major vascular structure (e.g. carotid artery)
* Tumor(s) in location that would potentially result in significant clinical adverse effects if post-treatment tumor swelling were to occur
* Clinically uncontrolled and/or rapidly accumulating ascites, pericardial and/or pleural effusions
* History of severe or unstable cardiac disease
* Current, known CNS malignancy (history of completely resected or irradiated brain metastases by WBRT or stereotactic radiosurgery allowed)
* Administered anti-cancer therapy within 4 weeks prior to first treatment (6 weeks in case of mitomycin C or nitrosoureas)
* Use of anti-viral, anti-platelet, or anti-coagulation medication [Patients who discontinue such medications within 7 days prior to first treatment may be eligible for this study.] Low dose aspirin (approximately 81 mg) allowed.
* Pulse oximetry O2 saturation <90% Pulse oximetry O2 saturation <90% at rest
* Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination
* Pregnant or nursing
* Household contact exclusions:
* Women who are pregnant or nursing an infant
* Children < 5 years old
* People with skin disease (e.g. eczema, atopic dermatitis, and related diseases
* Immunocompromised hosts (severe deficiencies in cell-mediated immunity, including AIDS, organ transplant recipients, hematologic malignancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximally-tolerated dose (MTD) and/or maximum-feasible dose (MFD) of JX-594 administered by biweekly intravenous (IV) infusion | DLT evaluations through 14 days following last JX-594 treatment
  Any of the following treatment related adverse events: Grade 4 toxicity, Grade 3 hematologic toxicity for > 5 days, Grade 3 non-hematologic toxicities persisting for > 7 days except for flu-like symptoms that respond to standard therapies.
Determine the safety of JX-594 administered by biweekly IV infusion | Safety evaluations through 28 days after last dose of JX-594
  Adverse events will be collected and assessed to assess safety and tolerability through 28 days after last dose of JX-594 (or until all events considered probably or possibly related to JX-594 have resolved, stabilized, or returned to baseline status).

SECONDARY OUTCOMES:
Determine the pharmacokinetics, pharmacodynamics and immune response activity of JX-594 | Blood samples collected at assigned time points from baseline through Week 8
  Change over time in viral genomes, infectious units, GM-CSF concentration, peripheral white blood cell counts, plasma cytokine measurements, and neutralizing antibodies to JX-594 in blood and/or serum.
Determine the anti-tumoral response of JX-594 | Disease control and response assessment at Week 8
  Tumor response (Stable, partial, complete, progression) by standard RECIST on CT/MRI. Decrease in tumor blood marker.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea